CLINICAL TRIAL: NCT00764478
Title: A Phase 3b, Multicenter, Double-Blind, Fixed-Dose, Parallel-Group, Three Week Placebo Controlled Trial Evaluating the Safety and Efficacy of Asenapine in Subjects With Bipolar 1 Disorder Experiencing an Acute Manic or Mixed Episode (Protocol P05691 [Formerly 041044])
Brief Title: Fixed-dose Safety and Efficacy Study of Asenapine for the Treatment of Acute Manic or Mixed Episode in Bipolar 1 Disorder (P05691)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05691; 2010-018409-13 (EudraCT Number); MK-8274-003 (Other: Merck)
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Results first posted 2015-04-24 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2022-02

CONDITIONS: Bipolar 1 Disorder
MeSH Terms: interventions — asenapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Asenapine 5 mg BID (Experimental): Participants were administered one 5 mg asenapine tablet, sublingually BID for 21 days
  Interventions: Drug: Asenapine
- Asenapine 10 mg BID (Experimental): Participants were administered one 10 mg asenapine tablet, sublingually BID for 21 days
  Interventions: Drug: Asenapine
- Placebo BID (Placebo Comparator): Participants were administered one asenapine-matched placebo tablet sublingually BID for 21 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asenapine — asenapine tablet, 5 mg sublingually BID for 21 days
  Other Names: SCH 900274, Saphris®, Sycrest®, Org 5222
  Arms: Asenapine 5 mg BID
Drug: Asenapine — asenapine tablet, 10 mg sublingually BID for 21 days
  Other Names: SCH 900274, Saphris®, Sycrest®, Org 5222
  Arms: Asenapine 10 mg BID
Drug: Placebo — placebo sublingual tablet, administered BID for 21 days
  Arms: Placebo BID

SUMMARY:
This trial will study the efficacy and safety of a fixed dose of asenapine in participants diagnosed with Bipolar 1 Disorder. Participants who qualify for the study will be randomly assigned to receive a fixed dose of asenapine (either 5 mg or 10 mg twice daily [BID]) or placebo (BID) for 3 weeks. Throughout the trial, observations will be made on each participant at various times to assess the safety and effectiveness of the study treatment. The primary hypothesis is that there is at least one dose of asenapine that is superior to placebo in the change from baseline in manic symptoms (as measured by Young Mania Rating Scale [YMRS]) at Day 21 of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Each participant must be at least 18 years of age
* Male, or a female who is not of child-bearing potential or who is non-pregnant, non-lactating, and is using a medically accepted method of contraception
* Each participant must have a current diagnosis of Bipolar I Disorder, current episode manic or mixed
* Each participant must be confirmed to be experiencing an acute manic or mixed bipolar 1 episode
* Each participant must have discontinued the use of all prohibited psychotropic medications

Exclusion Criteria:

* A participant must not have a primary Axis I disorder other than Bipolar 1 Disorder (i.e., an Axis 1 disorder other than Bipolar 1 Disorder that is primarily responsible for current symptoms and functional impairment)
* A participant must not currently (within the past 6 months) meet the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR™) criteria for substance abuse or dependence (excluding nicotine)
* A participant must not be at imminent risk of self-harm or harm to others, in the investigator's opinion based on clinical interview and responses provided on the Columbia Suicide Severity Rating Scale (CSSRS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2012-04-06 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2014-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Landbloom RL, Mackle M, Wu X, Kelly L, Snow-Adami L, McIntyre RS, Mathews M, Hundt C. Asenapine: Efficacy and safety of 5 and 10mg bid in a 3-week, randomized, double-blind, placebo-controlled trial in adults with a manic or mixed episode associated with bipolar I disorder. J Affect Disord. 2016 Jan 15;190:103-110. doi: 10.1016/j.jad.2015.06.059. Epub 2015 Sep 25. PMID 26496015

RESULTS

PARTICIPANT FLOW:
Groups:
- Asenapine 5 mg BID: Participants were administered one 5 mg asenapine tablet, sublingually twice daily (BID) for 21 days
Period: Overall Study
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Started | 122 | 119 | 126
Completed | 107 | 97 | 118
Not Completed | 15 | 22 | 8
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Withdrawal by Subject | 7 | 12 | 1
Not completed — Lost to Follow-up | 7 | 8 | 5
Not completed — Protocol Violation | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized participants who received at least one dose of trial medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID | Total
Number analyzed (Participants) | 122 | 119 | 126 | 367
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.3 (10.82) | 42.5 (11.06) | 44.6 (11.54) | 43.8 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 64 | 72 | 201
  Male | 57 | 55 | 54 | 166

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Young Mania Rating Scale (Y-MRS) Total Score at Day 21
Description: Y-MRS consists of responses to the following 11 items: elevated mood, increased motor activity energy, sexual interest, sleep, language-thought disorder, appearance, insight, irritability, speech - rate and amount, content and disruptive-aggressive behavior. The scores from the 11 items are summed to give a total score ranging from 0 to 60, with a higher score indicating greater severity of symptoms. The analysis is based on a mixed model repeated measures (MMRM) model. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 21
Population: Randomized participants who received at least one dose of trial medication and had at least one baseline and post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 120 | 113 | 126
Score on a scale | -14.4 (1.02) | -14.9 (1.04) | -10.9 (0.99)
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.0136, MMRM — Adjusted p-value from graphical approach to control Type 1 error rate among primary and secondary hypotheses; Least Square (LS) means difference = -3.5, 95% CI 2-sided [-6.3 to -0.7], Standard Error of Mean 1.41 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.0100, MMRM — Adjusted p-value from graphical approach to control Type 1 error rate among primary and secondary hypotheses; LS means difference = -4.0, 95% CI 2-sided [-6.9 to -1.2], Standard Error of Mean 1.43 — Asenapine 10 mg BID minus Placebo BID

2. Secondary Outcome: Change From Baseline in Clinical Global Impression - Bipolar Mania - Severity of Illness (CGI-BP-S) Overall Score at Day 21
Description: The CGI-BP-S is a score that measures the severity of overall bipolar illness. The score ranges on a scale from 1 to 7, where 1 is normal, and 7 is very severely ill. The analysis is based on a MMRM model. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 21
Population: Randomized participants who received at least one dose of trial medication and had at least one baseline and post-baseline measurement. One participant from the Placebo BID arm missed a baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 120 | 113 | 125
Score on a scale | -1.6 (0.12) | -1.7 (0.12) | -1.1 (0.11)
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.0100, MMRM — Adjusted p-value from Hochberg's method for testing two secondary efficacy hypotheses; LS means difference = -0.5, 95% CI 2-sided [-0.8 to -0.2], Standard Error of Mean 0.16 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.0052, MMRM — Adjusted p-value from Hochberg's method for testing two secondary efficacy hypotheses; LS means difference = -0.5, 95% CI 2-sided [-0.9 to -0.2], Standard Error of Mean 0.16 — Asenapine 10 mg BID minus Placebo BID

3. Secondary Outcome: Percentage of Participants Who Are Y-MRS Responders at Day 21
Description: Y-MRS consists of responses to the following 11 items: elevated mood, increased motor activity energy, sexual interest, sleep, language-thought disorder, appearance, insight, irritability, speech - rate and amount, content and disruptive-aggressive behavior. The scores from the 11 items are summed to give a total score ranging from 0 to 60, with a higher score indicating greater severity of symptoms. Missing data were imputed by Last Observation Carried Forward (LOCF). Y-MRS responders are defined as having a >= 50% decrease from baseline in Y-MRS total score.
Time Frame: Day 21
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 120 | 113 | 126
Percentage of participants | 45.0 | 46.9 | 39.7
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.5352, Cochran-Mantel-Haenszel — Overall adjusted p-value from Hochberg's method for testing two secondary efficacy hypotheses
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.4274, Cochran-Mantel-Haenszel — Overall adjusted p-value from Hochberg's method for testing two secondary efficacy hypotheses

4. Secondary Outcome: Change From Baseline in Y-MRS Total Score at Day 2, Day 4, Day 7 and Day 14
Description: Y-MRS consists of responses to the following 11 items: elevated mood, increased motor activity energy, sexual interest, sleep, language-thought disorder, appearance, insight, irritability, speech - rate and amount, content and disruptive-aggressive behavior. The scores from the 11 items are summed to give a total score ranging from 0 to 60, with a higher score indicating greater severity of symptoms. The analysis is based on a MMRM model. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 2, Day 4, Day 7 and Day 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 120 | 113 | 126
Score on a scale
  Day 2 | -5.6 (0.57) | -5.8 (0.59) | -2.9 (0.56)
  Day 4 | -8.6 (0.67) | -8.6 (0.68) | -4.9 (0.64)
  Day 7 | -10.0 (0.81) | -10.7 (0.83) | -6.6 (0.79)
  Day 14 | -11.1 (0.98) | -12.5 (1.00) | -9.4 (0.95)
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 2; Test type: Superiority or Other; p = 0.0007, MMRM; Least Square (LS) means difference = -2.7, 95% CI 2-sided [-4.2 to -1.1], Standard Error of Mean 0.78 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 2; Test type: Superiority or Other; p = 0.0003, MMRM; LS means difference = -2.9, 95% CI 2-sided [-4.4 to -1.3], Standard Error of Mean 0.79 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p < 0.0001, MMRM; LS means difference = -3.6, 95% CI 2-sided [-5.4 to -1.8], Standard Error of Mean 0.91 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p < 0.0001, MMRM; LS means difference = -3.7, 95% CI 2-sided [-5.5 to -1.9], Standard Error of Mean 0.92 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0021, MMRM; LS means difference = -3.5, 95% CI 2-sided [-5.7 to -1.3], Standard Error of Mean 1.12 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0002, MMRM; LS means difference = -4.2, 95% CI 2-sided [-6.4 to -2.0], Standard Error of Mean 1.13 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 7: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.1907, MMRM; LS means difference = -1.8, 95% CI 2-sided [-4.4 to 0.9], Standard Error of Mean 1.35 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 8: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0238, MMRM; LS means difference = -3.1, 95% CI 2-sided [-5.8 to -0.4], Standard Error of Mean 1.37 — Asenapine 10 mg BID minus Placebo BID

5. Secondary Outcome: Percentage of Participants Who Are Y-MRS Responders at Day 2, Day 4, Day 7, Day 14
Description: Y-MRS consists of responses to the following 11 items: elevated mood, increased motor activity energy, sexual interest, sleep, language-thought disorder, appearance, insight, irritability, speech - rate and amount, content and disruptive-aggressive behavior. The scores from the 11 items are summed to give a total score ranging from 0 to 60, with a higher score indicating greater severity of symptoms. Missing data were imputed by LOCF. Y-MRS responders are defined as having a >= 50% decrease from baseline in Y-MRS total score.
Time Frame: Day 2, Day 4, Day 7, Day 14
Population: Randomized participants who received at least one dose of trial medication and had at least one baseline and post-baseline measurement, and had evaluable post-baseline measurement at timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 120 | 113 | 126
Percentage of participants
  Day 2 (n = 117,111,123) | 12.0 | 14.4 | 8.9
  Day 4 (n = 120,113,126) | 21.7 | 23.0 | 8.7
  Day 7 (n = 120,113,126) | 31.7 | 28.3 | 19.8
  Day 14 (n = 120,113,126) | 36.7 | 40.7 | 33.3
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 2; Test type: Superiority or Other; p = 0.2922, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 2; Test type: Superiority or Other; p = 0.1001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.0011, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.0011, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0194, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0841, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.4858, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.2496, Cochran-Mantel-Haenszel

6. Secondary Outcome: Percentage of Participants Who Are Y-MRS Remitters at Day 21
Description: Y-MRS consists of responses to the following 11 items: elevated mood, increased motor activity energy, sexual interest, sleep, language-thought disorder, appearance, insight, irritability, speech - rate and amount, content and disruptive-aggressive behavior. The 11 items are summed to give a total score ranging from 0 to 60, with a higher score indicating greater severity of symptoms. Missing data were imputed by LOCF. Y-MRS remitters are defined as having a Y-MRS total score of 12 or lower.
Time Frame: Day 21
Population: Randomized participants who received at least one dose of trial medication and had at least one post-baseline measurement.
Measure: Number; unit: Percentage of participants
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 120 | 113 | 126
Percentage of participants | 34.2 | 38.1 | 30.2
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.2912, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.1151, Cochran-Mantel-Haenszel

7. Secondary Outcome: Percentage of Participants Who Are Y-MRS Remitters at Day 2, Day 4, Day 7, Day 14, Day 21
Description: Y-MRS consists of responses to the following 11 items: elevated mood, increased motor activity energy, sexual interest, sleep, language-thought disorder, appearance, insight, irritability, speech - rate and amount, content and disruptive-aggressive behavior. The scores from the 11 items are summed to give a total score ranging from 0 to 60, with a higher score indicating greater severity of symptoms. The analysis is based on a generalized linear mixed model (GLMM). Y-MRS remitters are defined as having a Y-MRS total score of 12 or lower.
Time Frame: Day 2, Day 4, Day 7, Day 14, Day 21
Population: Randomized participants who received at least one dose of trial medication and had at least one post-baseline measurement, and had evaluable post-baseline measurement at timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 120 | 113 | 126
Percentage of participants
  Day 2 (n= 117,111, 123) | 8.5 | 11.7 | 5.7
  Day 4 (n= 104, 106,118) | 17.3 | 15.1 | 10.2
  Day 7 (n= 104, 101,110) | 26.9 | 24.8 | 17.3
  Day 14 (n= 96, 91,102) | 28.1 | 27.5 | 24.5
  Day 21 (n= 86, 83,93) | 40.7 | 43.4 | 34.4

8. Secondary Outcome: Change From Baseline in Montgomery Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS measures depression and consists of 10 items, each rated on a scale from 0 to 6. The MADRS total score sums the scores from the 10 items, ranging from 0 to 60, with a higher numeric rating implying a greater degree of symptom severity. Missing data were imputed by LOCF. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 7 and Day 21
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 115 | 110 | 123
Score on a scale
  Day 7 (n=112,106, 117) | -4.3 (0.47) | -4.2 (0.48) | -2.3 (0.46)
  Day 21 (n =115, 110,123) | -4.6 (0.61) | -5.1 (0.63) | -2.5 (0.60)
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0019, ANCOVA
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0045, ANCOVA
Statistical Analysis 3: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0112, ANCOVA
Statistical Analysis 4: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0021, ANCOVA

9. Secondary Outcome: Change From Baseline in CGI-BP-S Overall Score at Day 2, Day 4, Day 7, Day 14
Description: as for outcome 2
Time Frame: Baseline and Day 2, Day 4, Day 7, Day 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 120 | 113 | 125
Score on a scale
  Day 2 | -0.5 (0.05) | -0.4 (0.06) | -0.2 (0.05)
  Day 4 | -0.8 (0.07) | -0.7 (0.07) | -0.4 (0.07)
  Day 7 | -1.0 (0.09) | -1.1 (0.09) | -0.7 (0.09)
  Day 14 | -1.3 (0.10) | -1.3 (0.11) | -1.0 (0.10)
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 2; Test type: Superiority or Other; p < 0.0001, MMRM; LS means difference = -0.3, 95% CI 2-sided [-0.4 to -0.1], Standard Error of Mean 0.07 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 2; Test type: Superiority or Other; p = 0.0076, MMRM; LS means difference = -0.2, 95% CI 2-sided [-0.3 to -0.1], Standard Error of Mean 0.07 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.0004, MMRM; LS means difference = -0.4, 95% CI 2-sided [-0.6 to -0.2], Standard Error of Mean 0.10 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.0040, MMRM; LS means difference = -0.3, 95% CI 2-sided [-0.5 to -0.1], Standard Error of Mean 0.10 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0061, MMRM; LS means difference = -0.3, 95% CI 2-sided [-0.6 to -0.1], Standard Error of Mean 0.12 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0031, MMRM; LS means difference = -0.4, 95% CI 2-sided [-0.6 to -0.1], Standard Error of Mean 0.13 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 7: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.1086, MMRM; LS means difference = -0.2, 95% CI 2-sided [-0.5 to 0.1], Standard Error of Mean 0.14 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 8: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0376, MMRM; LS means difference = -0.3, 95% CI 2-sided [-0.6 to -0.0], Standard Error of Mean 0.15 — Asenapine 10 mg BID minus Placebo BID

10. Secondary Outcome: Change From Baseline in CGI-BP-S Mania Score
Description: The CGI-BP-S mania is a score that assesses the severity of the mania component of bipolar illness. The score ranges on a scale from 1 to 7, where 1 is normal, and 7 is very severely ill. Missing data were imputed by LOCF. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 2, Day 4, Day 7, Day 14, and Day 21
Population: Randomized participants who received at least one dose of trial medication and had at least one baseline and post-baseline measurement, and had evaluable post-baseline measurement at timepoint. One participant from the Placebo BID arm missed a baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 120 | 113 | 125
Score on a scale
  Day 2 (n=118,111,122) | -0.4 (0.06) | -0.4 (0.06) | -0.1 (0.06)
  Day 4 (n=120,113,125) | -0.7 (0.07) | -0.7 (0.08) | -0.3 (0.07)
  Day 7 (n=120,113,125) | -0.9 (0.09) | -1.0 (0.09) | -0.7 (0.09)
  Day 14 (n=120,113,125) | -1.2 (0.10) | -1.3 (0.11) | -1.0 (0.10)
  Day 21 (n=120,113,125) | -1.4 (0.11) | -1.5 (0.12) | -1.1 (0.11)
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 2; Test type: Superiority or Other; p = 0.0005, ANCOVA
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 2; Test type: Superiority or Other; p = 0.0026, ANCOVA
Statistical Analysis 3: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.0007, ANCOVA
Statistical Analysis 4: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.0002, ANCOVA
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0387, ANCOVA
Statistical Analysis 6: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0059, ANCOVA
Statistical Analysis 7: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.3110, ANCOVA
Statistical Analysis 8: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0613, ANCOVA
Statistical Analysis 9: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0640, ANCOVA
Statistical Analysis 10: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0139, ANCOVA

11. Secondary Outcome: Change From Baseline in CGI-BP-S Depression Score
Description: The CGI-BP-S depression is a score that assesses the severity of the depression component of bipolar illness. The score ranges on a scale from 1 to 7, where 1 is normal, and 7 is very severely ill. Missing data were imputed by LOCF. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 2, Day 4, Day 7, Day 14, and Day 21
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 120 | 113 | 125
Score on a scale
  Day 2 (n=118,111,122) | -0.2 (0.06) | -0.2 (0.06) | -0.2 (0.06)
  Day 4 (n=120,113,125) | -0.3 (0.06) | -0.3 (0.06) | -0.3 (0.06)
  Day 7 (n=120,113,125) | -0.3 (0.07) | -0.4 (0.07) | -0.1 (0.07)
  Day 14 (n=120,113,125) | -0.4 (0.07) | -0.5 (0.07) | -0.2 (0.07)
  Day 21 (n=120,113,125) | -0.4 (0.08) | -0.5 (0.08) | -0.1 (0.08)
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 2; Test type: Superiority or Other; p = 0.9708, ANCOVA
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 2; Test type: Superiority or Other; p = 0.7891, ANCOVA
Statistical Analysis 3: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.5222, ANCOVA
Statistical Analysis 4: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.8686, ANCOVA
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0696, ANCOVA
Statistical Analysis 6: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0049, ANCOVA
Statistical Analysis 7: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0196, ANCOVA
Statistical Analysis 8: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0032, ANCOVA
Statistical Analysis 9: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0061, ANCOVA
Statistical Analysis 10: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0012, ANCOVA

12. Secondary Outcome: Percentage of Participants Who Are CGI-BP Improvement (CGI-BP-I) Responders of Overall Bipolar Illness Score
Description: The CGI-BP-I overall is a score on a 7-point scale for assessing the change from preceding phase of overall symptoms of bipolar disorder during the treatment of an acute episode or in longer term illness prophylaxis. Compared to the baseline, the CGI-BP-I overall score ranges from 1 = very much improved since initiating treatment, to 7 = very much worse since initiating treatment. Missing data were imputed by LOCF. A CGI-BP-I responder had a score of 3 (minimally improved) or lower.
Time Frame: Day 2, Day 4, Day 7, Day 14, and Day 21
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 120 | 113 | 126
Percentage of participants
  Day 2 (n=118,111,123) | 50.8 | 45.9 | 37.4
  Day 4 (n=120,113,126) | 64.2 | 64.6 | 55.6
  Day 7 (n=120,113,126) | 73.3 | 78.8 | 61.1
  Day 14 (n=120,113,126) | 70.8 | 83.2 | 65.1
  Day 21 (n=120,113,126) | 74.2 | 82.3 | 64.3
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 2; Test type: Superiority or Other; p = 0.0147, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 2; Test type: Superiority or Other; p = 0.0720, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.1213, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.0588, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0200, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0017, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.2401, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0009, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0525, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0025, Cochran-Mantel-Haenszel

13. Secondary Outcome: Percentage of Participants Who Are CGI-BP Improvement (CGI-BP-I) Responders of Mania Score
Description: The CGI-BP-I mania is a score on a 7-point scale for assessing the change from preceding phase of mania symptoms of bipolar disorder during the treatment of an acute episode or in longer term illness prophylaxis. Compared to the baseline, the CGI-BP-I mania score ranges from 1 = very much improved since initiating treatment, to 7 = very much worse since initiating treatment. Missing data were imputed by LOCF. A CGI-BP-I responder had a score of 3 (minimally improved) or lower.
Time Frame: Day 2, Day 4, Day 7, Day 14, and Day 21
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 120 | 113 | 126
Percentage of participants
  Day 2 (n=118,111,123) | 49.2 | 45.9 | 37.4
  Day 4 (n=120,113,126) | 64.2 | 66.4 | 55.6
  Day 7 (n=120,113,126) | 74.2 | 80.5 | 63.5
  Day 14 (n=120,113,126) | 75.8 | 82.3 | 66.7
  Day 21 (n=120,113,126) | 79.2 | 84.1 | 66.7
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 2; Test type: Superiority or Other; p = 0.0377, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 2; Test type: Superiority or Other; p = 0.0771, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.1264, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.0280, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0583, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0021, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0866, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0048, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0147, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0030, Cochran-Mantel-Haenszel

14. Secondary Outcome: Percentage of Participants Who Are CGI-BP Improvement (CGI-BP-I) Responders of Depression Score
Description: The CGI-BP-I depression is a score on a 7-point scale for assessing the change from preceding phase of depression symptoms of bipolar disorder during the treatment of an acute episode or in longer term illness prophylaxis. Compared to the baseline, the CGI-BP-I depression score ranges from 1 = very much improved since initiating treatment, to 7 = very much worse since initiating treatment. Missing data were imputed by LOCF. A CGI-BP-I responder had a score of 3 (minimally improved) or lower.
Time Frame: Day 2, Day 4, Day 7, Day 14, and Day 21
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 117 | 106 | 121
Percentage of participants
  Day 2 (n=113, 103, 116) | 21.2 | 28.2 | 11.2
  Day 4 (n=116, 106, 119) | 26.7 | 32.1 | 19.3
  Day 7 (n=117, 106, 119) | 31.6 | 35.8 | 23.5
  Day 14 (n=117, 106, 120) | 31.6 | 42.5 | 26.7
  Day 21 (n=117, 106, 121) | 32.5 | 44.3 | 28.9
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 2; Test type: Superiority or Other; p = 0.0104, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 2; Test type: Superiority or Other; p = 0.0005, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.0692, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.0128, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0809, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0260, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.2576, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0077, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.3960, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0141, Cochran-Mantel-Haenszel

15. Secondary Outcome: Change From Baseline in Positive And Negative Syndrome Scale (PANSS) Total Score
Description: PANSS total score measures symptoms of schizophrenia and consists of responses to 30 items: 7 items from the positive subscale (P1-P7), 7 items from the negative subscale (N1-N7) and 16 items from the general psychopathology subscale (G1-G16). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS total score sums the scores from all 30 items, and ranges from 30 to 210, with a higher score indicating greater severity of symptoms. The analysis is based on a MMRM model. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 7, Day 14, Day 21
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 115 | 110 | 123
Score on a scale
  Day 7 | -6.9 (0.77) | -6.9 (0.79) | -3.9 (0.76)
  Day 14 | -7.5 (0.96) | -8.4 (0.99) | -5.2 (0.94)
  Day 21 | -9.3 (1.02) | -8.8 (1.05) | -5.5 (1.00)
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0056, MMRM; Least Square (LS) means difference = -3.0, 95% CI 2-sided [-5.1 to -0.9], Standard Error of Mean 1.06 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0068, MMRM; LS means difference = -2.9, 95% CI 2-sided [-5.0 to -0.8], Standard Error of Mean 1.08 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0743, MMRM; LS means difference = -2.4, 95% CI 2-sided [-5.0 to 0.2], Standard Error of Mean 1.33 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0177, MMRM; LS means difference = -3.2, 95% CI 2-sided [-5.9 to -0.6], Standard Error of Mean 1.35 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0081, MMRM; LS means difference = -3.8, 95% CI 2-sided [-6.6 to -1.0], Standard Error of Mean 1.41 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0247, MMRM; LS means difference = -3.2, 95% CI 2-sided [-6.1 to -0.4], Standard Error of Mean 1.43 — Asenapine 10 mg BID minus Placebo BID

16. Secondary Outcome: Change From Baseline in PANSS Negative Subscale Score
Description: PANSS Negative subscale measures symptoms of schizophrenia and consists of responses to 7 items (N1-N7). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS Negative subscale sums the scores from all 7 items and ranges from 7 to 49, with a higher score indicating greater severity of symptoms. The analysis is based on a MMRM model. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 7, Day 14, Day 21
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 115 | 110 | 123
Score on a scale
  Day 7 | -0.5 (0.22) | -0.8 (0.22) | -0.5 (0.21)
  Day 14 | -0.8 (0.23) | -0.7 (0.24) | -0.8 (0.23)
  Day 21 | -0.4 (0.28) | -0.0 (0.29) | -0.4 (0.27)
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.9808, MMRM; Least Square (LS) means difference = -0.0, 95% CI 2-sided [-0.6 to 0.6], Standard Error of Mean 0.30 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.2830, MMRM; LS means difference = -0.3, 95% CI 2-sided [-0.9 to 0.3], Standard Error of Mean 0.31 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.9751, MMRM; LS means difference = -0.0, 95% CI 2-sided [-0.6 to 0.6], Standard Error of Mean 0.32 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.7879, MMRM; LS means difference = 0.1, 95% CI 2-sided [-0.6 to 0.7], Standard Error of Mean 0.33 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.9654, MMRM; LS means difference = -0.0, 95% CI 2-sided [-0.8 to 0.7], Standard Error of Mean 0.38 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.3917, MMRM; LS means difference = 0.3, 95% CI 2-sided [-0.4 to 1.1], Standard Error of Mean 0.39 — Asenapine 10 mg BID minus Placebo BID

17. Secondary Outcome: Change From Baseline in PANSS Positive Subscale Score
Description: PANSS Positive subscale measures symptoms of schizophrenia and consists of responses to 7 items (P1-P7). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS Positive subscale sums the scores from all 7 items and ranges from 7 to 49, with a higher score indicating greater severity of symptoms. The analysis is based on a MMRM model. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 7, Day 14, Day 21
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 115 | 110 | 123
Score on a scale
  Day 7 | -2.4 (0.30) | -2.8 (0.31) | -1.4 (0.29)
  Day 14 | -2.3 (0.37) | -3.2 (0.38) | -2.1 (0.36)
  Day 21 | -3.5 (0.37) | -3.9 (0.38) | -2.4 (0.36)
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0120, MMRM; Least Square (LS) means difference = -1.0, 95% CI 2-sided [-1.8 to -0.2], Standard Error of Mean 0.41 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0011, MMRM; LS means difference = -1.4, 95% CI 2-sided [-2.2 to -0.5], Standard Error of Mean 0.42 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.6885, MMRM; LS means difference = -0.2, 95% CI 2-sided [-1.2 to 0.8], Standard Error of Mean 0.51 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0398, MMRM; LS means difference = -1.1, 95% CI 2-sided [-2.1 to -0.1], Standard Error of Mean 0.52 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0258, MMRM; LS means difference = -1.1, 95% CI 2-sided [-2.1 to -0.1], Standard Error of Mean 0.51 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0031, MMRM; LS means difference = -1.5, 95% CI 2-sided [-2.5 to -0.5], Standard Error of Mean 0.51 — Asenapine 10 mg BID minus Placebo BID

18. Secondary Outcome: Change From Baseline in PANSS General Psychopathology Subscale Score
Description: PANSS General Psychopathology subscale measures symptoms of schizophrenia and consists of responses to 16 items (G1-G16). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS General Psychopathology subscale sums the scores from all 16 items and ranges from 16 to 112, with a higher score indicating greater severity of symptoms. The analysis is based on a MMRM model. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 7, Day 14, Day 21
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 115 | 110 | 123
Score on a scale
  Day 7 | -4.0 (0.46) | -3.3 (0.48) | -2.1 (0.46)
  Day 14 | -4.5 (0.57) | -4.6 (0.59) | -2.4 (0.56)
  Day 21 | -5.5 (0.61) | -4.9 (0.62) | -2.9 (0.59)
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0033, MMRM; Least Square (LS) means difference = -1.9, 95% CI 2-sided [-3.2 to -0.6], Standard Error of Mean 0.64 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0622, MMRM; LS means difference = -1.2, 95% CI 2-sided [-2.5 to 0.1], Standard Error of Mean 0.65 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0083, MMRM; LS means difference = -2.1, 95% CI 2-sided [-3.6 to -0.5], Standard Error of Mean 0.79 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0064, MMRM; LS means difference = -2.2, 95% CI 2-sided [-3.8 to -0.6], Standard Error of Mean 0.80 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0022, MMRM; LS means difference = -2.6, 95% CI 2-sided [-4.3 to -0.9], Standard Error of Mean 0.84 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0196, MMRM; LS means difference = -2.0, 95% CI 2-sided [-3.7 to -0.3], Standard Error of Mean 0.85 — Asenapine 10 mg BID minus Placebo BID

19. Secondary Outcome: Change From Baseline in PANSS Marder Factor Positive Symptom Score
Description: PANSS Marder Factor Positive symptom score measures symptoms of schizophrenia and consists of responses to 8 items (P1,P3,P5,P6,N7,G1,G9,G12). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS Marder Factor Positive symptom score sums the scores from all 8 items and ranges from 8 to 56, with a higher score indicating greater severity of symptoms. The analysis is based on a MMRM model. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 7, Day 14, Day 21
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 115 | 110 | 123
Score on a scale
  Day 7 | -1.9 (0.29) | -1.9 (0.29) | -1.3 (0.28)
  Day 14 | -1.6 (0.33) | -2.5 (0.34) | -1.6 (0.33)
  Day 21 | -2.6 (0.34) | -2.9 (0.35) | -1.7 (0.33)
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.1883, MMRM; Least Square (LS) means difference = -0.5, 95% CI 2-sided [-1.3 to 0.3], Standard Error of Mean 0.40 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.1684, MMRM; LS means difference = -0.6, 95% CI 2-sided [-1.3 to 0.2], Standard Error of Mean 0.40 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.9522, MMRM; LS means difference = -0.0, 95% CI 2-sided [-0.9 to 0.9], Standard Error of Mean 0.46 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0514, MMRM; LS means difference = -0.9, 95% CI 2-sided [-1.8 to 0.0], Standard Error of Mean 0.47 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0531, MMRM; LS means difference = -0.9, 95% CI 2-sided [-1.8 to 0.0], Standard Error of Mean 0.47 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0078, MMRM; LS means difference = -1.3, 95% CI 2-sided [-2.2 to -0.3], Standard Error of Mean 0.48 — Asenapine 10 mg BID minus Placebo BID

20. Secondary Outcome: Change From Baseline in PANSS Marder Factor Negative Symptom Score
Description: PANSS Marder Factor Negative symptom score measures symptoms of schizophrenia and consists of responses to 7 items (N1,N2,N3,N4,N6,G7,G16). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS Marder Factor Negative symptom score sums the scores from all 7 items and ranges from 7 to 49, with a higher score indicating greater severity of symptoms. The analysis is based on a MMRM model. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 7, Day 14, Day 21
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 115 | 110 | 123
Score on a scale
  Day 7 | -0.5 (0.23) | -0.8 (0.24) | -0.5 (0.23)
  Day 14 | -0.6 (0.24) | -0.5 (0.25) | -0.7 (0.24)
  Day 21 | -0.1 (0.27) | 0.1 (0.28) | -0.1 (0.27)
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.7746, MMRM; Least Square (LS) means difference = -0.1, 95% CI 2-sided [-0.7 to 0.5], Standard Error of Mean 0.32 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.2754, MMRM; LS means difference = -0.4, 95% CI 2-sided [-1.0 to 0.3], Standard Error of Mean 0.32 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.9109, MMRM; LS means difference = 0.0, 95% CI 2-sided [-0.6 to 0.7], Standard Error of Mean 0.34 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.7295, MMRM; LS means difference = 0.1, 95% CI 2-sided [-0.6 to 0.8], Standard Error of Mean 0.34 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.9800, MMRM; LS means difference = 0.0, 95% CI 2-sided [-0.7 to 0.8], Standard Error of Mean 0.38 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.5122, MMRM; LS means difference = 0.3, 95% CI 2-sided [-0.5 to 1.0], Standard Error of Mean 0.38 — Asenapine 10 mg BID minus Placebo BID

21. Secondary Outcome: Change From Baseline in PANSS Marder Factor Disorganized Thought Symptom Score
Description: PANSS Marder Factor Disorganized Thought symptom score measures symptoms of schizophrenia and consists of responses to 7 items (P2,N5,G5,G10,G11,G13,G15). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS Marder Factor Disorganized Thought symptom score sums the scores from all 7 items and ranges from 7 to 49, with a higher score indicating greater severity of symptoms. The analysis is based on a MMRM model. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 7, Day 14, Day 21
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 115 | 110 | 123
Score on a scale
  Day 7 | -1.1 (0.21) | -1.3 (0.22) | -0.7 (0.21)
  Day 14 | -1.5 (0.26) | -1.8 (0.27) | -1.2 (0.26)
  Day 21 | -2.0 (0.28) | -1.7 (0.29) | -1.5 (0.27)
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.2191, MMRM; Least Square (LS) means difference = -0.4, 95% CI 2-sided [-0.9 to 0.2], Standard Error of Mean 0.29 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0589, MMRM; LS means difference = -0.6, 95% CI 2-sided [-1.1 to 0.0], Standard Error of Mean 0.29 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.3683, MMRM; LS means difference = -0.3, 95% CI 2-sided [-1.0 to 0.4], Standard Error of Mean 0.36 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0982, MMRM; LS means difference = -0.6, 95% CI 2-sided [-1.3 to 0.1], Standard Error of Mean 0.37 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.1969, MMRM; LS means difference = -0.5, 95% CI 2-sided [-1.3 to 0.3], Standard Error of Mean 0.38 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.5615, MMRM; LS means difference = -0.2, 95% CI 2-sided [-1.0 to 0.5], Standard Error of Mean 0.39 — Asenapine 10 mg BID minus Placebo BID

22. Secondary Outcome: Change From Baseline in PANSS Marder Factor Hostility/Excitement Symptom Score
Description: PANSS Marder Factor Hostility/Excitement symptom score measures symptoms of schizophrenia and consists of responses to 4 items (P4,P7,G8,G14). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS Marder Factor Hostility/Excitement symptom score sums the score from all 4 items and ranges from 4 to 28, with a higher score indicating greater severity of symptoms. The analysis is based on a MMRM model. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 7, Day 14, Day 21
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 115 | 110 | 123
Score on a scale
  Day 7 | -1.7 (0.24) | -1.7 (0.25) | -0.9 (0.24)
  Day 14 | -1.8 (0.28) | -2.0 (0.29) | -1.2 (0.27)
  Day 21 | -2.6 (0.29) | -2.5 (0.30) | -1.5 (0.28)
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0101, MMRM; Least Square (LS) means difference = -0.9, 95% CI 2-sided [-1.5 to -0.2], Standard Error of Mean 0.33 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0146, MMRM; LS means difference = -0.8, 95% CI 2-sided [-1.5 to -0.2], Standard Error of Mean 0.34 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0861, MMRM; LS means difference = -0.7, 95% CI 2-sided [-1.4 to 0.1], Standard Error of Mean 0.39 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0342, MMRM; LS means difference = -0.8, 95% CI 2-sided [-1.6 to -0.1], Standard Error of Mean 0.39 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0037, MMRM; LS means difference = -1.2, 95% CI 2-sided [-2.0 to -0.4], Standard Error of Mean 0.40 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0096, MMRM; LS means difference = -1.1, 95% CI 2-sided [-1.9 to -0.3], Standard Error of Mean 0.41 — Asenapine 10 mg BID minus Placebo BID

23. Secondary Outcome: Change From Baseline in PANSS Marder Factor Anxiety/Depression Symptom Score
Description: PANSS Marder Factor Anxiety/Depression symptom score measures symptoms of schizophrenia and consists of responses to 4 items (G2,G3,G4,G6). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS Marder Factor Anxiety/Depression symptom score sums the scores from all 4 items and ranges from 4 to 28, with a higher score indicating greater severity of symptoms. The analysis is based on a MMRM model. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 7, Day14, Day 21
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 115 | 110 | 123
Score on a scale
  Day 7 | -1.7 (0.24) | -1.3 (0.24) | -0.7 (0.23)
  Day 14 | -2.0 (0.26) | -1.7 (0.27) | -0.7 (0.26)
  Day 21 | -2.1 (0.30) | -1.9 (0.30) | -1.0 (0.29)
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0019, MMRM; Least Square (LS) means difference = -1.0, 95% CI 2-sided [-1.7 to -0.4], Standard Error of Mean 0.32 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.0791, MMRM; LS means difference = -0.6, 95% CI 2-sided [-1.2 to 0.1], Standard Error of Mean 0.33 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0006, MMRM; LS means difference = -1.2, 95% CI 2-sided [-2.0 to -0.5], Standard Error of Mean 0.36 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0123, MMRM; LS means difference = -0.9, 95% CI 2-sided [-1.6 to -0.2], Standard Error of Mean 0.37 — Asenapine 10 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0054, MMRM; LS means difference = -1.1, 95% CI 2-sided [-2.0 to -0.3], Standard Error of Mean 0.41 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Asenapine 10 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0350, MMRM; LS means difference = -0.9, 95% CI 2-sided [-1.7 to -0.1], Standard Error of Mean 0.41 — Asenapine 10 mg BID minus Placebo BID

ADVERSE EVENTS:
Time Frame: Up to 33 days after end of treatment (up to 54 days)
Description: Randomized participants who received at least one dose of trial medication
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Serious Adverse Events (participants affected / at risk) | 3/122 | 1/119 | 2/126
Other Adverse Events (participants affected / at risk) | 43/122 | 67/119 | 24/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine 5 mg BID (N=122) | Asenapine 10 mg BID (N=119) | Placebo BID (N=126)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine 5 mg BID (N=122) | Asenapine 10 mg BID (N=119) | Placebo BID (N=126)
Hypoaesthesia oral (Gastrointestinal disorders) | 15 (15) | 27 (28) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 6 (6) | 4 (6)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 7 (7) | 3 (3)
Akathisia (Nervous system disorders) | 5 (5) | 18 (25) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5) | 6 (6) | 6 (6)
Dysgeusia (Nervous system disorders) | 4 (4) | 11 (11) | 0 (0)
Headache (Nervous system disorders) | 9 (10) | 6 (7) | 9 (11)
Sedation (Nervous system disorders) | 12 (12) | 18 (19) | 2 (2)
Somnolence (Nervous system disorders) | 12 (12) | 14 (15) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days to submission for publication or presentation, review copies of abstracts or manuscripts for publication (including without limitation, slides and texts of oral or other public presentations and texts of any transmission through any electronic media, eg, any computer access system such as the Internet, World Wide Web, etc) that report any results of the trial.